CLINICAL TRIAL: NCT05398198
Title: A Randomized, Double-blind, Placebo Controlled, Repeat Dose Phase 1b Study to Assess the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled GSK3923868 During Experimental Human Rhinovirus Infection in Participants With Mild Asthma
Brief Title: Efficacy and Safety of GSK3923868 Inhalation Powder, During Experimental Human Rhinovirus Infection in Participants With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213499; 2021-006640-27 (EudraCT Number)
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK3923868; Chronic Obstructive Pulmonary Disease (COPD); Respiratory Tract Diseases; Respiration Disorders; Pharmacokinetics; Pharmacodynamics; Human Rhinovirus (HRV); Viral Challenge
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Part A: In therapeutic treatment cohorts (cohort 1 and 2) repeat doses of GSK3923868 are administered after experimental viral infection with increasing time windows between viral inoculation and the initiation of study drug. The treatment is initiated 2, 3 and 4 days post-viral inoculation for cohort 1 and 2.
  Part B: In prophylactic treatment cohort (cohort 3), treatment is initiated before inoculation with virus.
  Of 3 cohorts planned, two cohorts will be performed (Cohort 1 and either Cohort 2 or 3). Cohort 1 data will be used to determine which cohort to progress to along with any study design changes.
Who Masked: Participant, Investigator
Masking Description: The participants and site staff will be blinded to the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GSK3923868 (Experimental): All participants in this arm will receive GSK3923868
  Interventions: Drug: GSK3923868
- Placebo (Placebo Comparator): All participants in this arm will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3923868 — GSK3923868 dose and administration as per study intervention.
  Arms: GSK3923868
Drug: Placebo — Placebo matching GSK3923868 will be administered.
  Arms: Placebo

SUMMARY:
This is a Phase 1b, single center study designed to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GSK3923868 following repeat doses in mild asthmatics during experimental human rhinovirus 16 (HRV-16) infection. The study will be conducted in two parts. Part A will determine the efficacy of GSK3923868 administration after viral inoculation (i.e., therapeutic treatment) and Part B may be undertaken to determine the efficacy of GSK3923868 administration before viral inoculation (i.e., prophylactic treatment). The purpose of this study is to establish proof-of-mechanism that GSK3923868 treatment can reduce symptoms of Human Rhinovirus (HRV) infection in a controlled setting.

ELIGIBILITY:
Inclusion Criteria:

* All Participant aged between 18 to 65 years of age (inclusive).
* Participants with a diagnosis of asthma.
* A screening pre-bronchodilator FEV1 greater than or equal to (≥) 65 percentage (%) predicted normal value.
* Positive Methacholine challenge test, defined as ≥ 20% fall in FEV1 at a methacholine concentration less than or equal to (≤) 16 milligram/milliliter (mg/mL) at Screening.

If the methacholine challenge test is negative or the participant is unable to perform this test, bronchodilator reversibility is allowed as an alternative, assessed as follows:

* Positive bronchodilator reversibility test, defined as an increase in FEV1 >12% and >200 mL from baseline, 10 to 15 minutes after administration of 400 micrograms (mcg) salbutamol (or equivalent).
* Participants with positive skin prick test.
* The HRV-16 neutralization antibody assay indicates that the participant will be susceptible to HRV-16 infection.
* Participants with controlled asthma, using short-acting beta agonist (SABA) or intermittent inhaled corticosteroid (ICS) or ICS/ long-acting beta agonist (LABA) therapy.
* Male and female- A female participant is eligible to participate if she is not pregnant or breastfeeding.
* Participant capable of giving signed informed consent.

Exclusion Criteria:

All participants:

* Any asthma exacerbation requiring systemic corticosteroids within 8 weeks of admission, or that resulted in overnight hospitalization requiring additional treatment for asthma within 3 months of admission.
* History of life-threatening asthma, defined as any asthma episode that required admission to a high-dependency or intensive therapy unit.
* The presence of concurrent significant pulmonary diseases, other than asthma, including bronchiectasis, pulmonary fibrosis, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other significant respiratory abnormalities.
* Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the study.
* Any clinically significant history of epistaxis (large nosebleeds) within the last 3 months of admission and/or history of being hospitalized due to epistaxis on any previous occasion.
* Any nasal or sinus surgery within 3 months of admission with any acute illness, including a common cold or other respiratory tract infection within 6 weeks before admission.
* Any major illness or hospitalization within 6 months before admission to the unit.
* Lifetime history of anaphylaxis or severe allergic reaction or significant intolerance to any food or drug.
* Fridericia's QT correction formula (QTcF) >450 millisecond (msec) on Day -1 based on the average of triplicate ECGs.
* Evidence of vaccinations within the 4 weeks prior to the planned date of viral challenge.
* Intention to receive any vaccination before the last day of follow up.
* Prior participation in another Human Viral Challenge study with a respiratory virus in the preceding 12 months.
* Positive pathogen screen for respiratory tract infection
* History of regular use of tobacco or nicotine-containing products.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that contraindicates participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) of change from baseline (CfB) in total lower respiratory tract symptoms (LRTS) score from day of inoculation up to discharge | Baseline and up to Day 15
  The LRTS includes cough, chest tightness, shortness of breath, wheezing, daily activity, and night time awakenings. Each symptom is assessed on a 4-point scale. The score ranges from 0 to 3, where higher points indicate more symptoms experienced and severity that restricts normal activities. Shortness of breath and wheezing will be measured on a 5-point scale and ranges from 0 to 4 in which 0 indicates no symptoms and 4 indicates symptoms at total rest and the highest level of disease severity. LRTS assessment is performed three times a day.

SECONDARY OUTCOMES:
Maximal CfB in total LRTS score from day of inoculation up to discharge | Baseline and up to Day 15
AUC and maximal CfB in total upper respiratory tract symptoms (URTS) score from day of inoculation up to discharge | Baseline and up to Day 15
  The URTS includes nasal discharge, nasal obstruction, sneezing and sore throat. Each symptom will be assessed on a 4-point scale, where 0 indicates no symptom and a higher point for more symptoms and severity that restricts normal activities.
Mean percent CfB and maximum percent decline from baseline in trough force expiratory volume (FEV1) from day of inoculation up to discharge | Baseline and up to Day 15
Mean percent CfB and maximum percent decline from baseline in morning and evening peak expiratory flow (PEF) from day of inoculation up to discharge | Baseline and up to Day 15
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 22
Number of participants with clinically significant changes in vital signs | Up to Day 22
Number of participants with clinically significant changes in electrocardiogram (ECG) | Up to Day 22
Number of participants with clinically significant changes in clinical laboratory parameters | Up to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com